CLINICAL TRIAL: NCT01674426
Title: Pathogenesis of Functional Hypothalamic Amenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Sarah Berga, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MH50748
Record Dates: First submitted 2012-08-14; First posted 2012-08-28 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Disorder of Endocrine Ovary; Hypersecretion; Cortisol; Metabolic Disturbance; Stress, Psychological
Keywords: functional hypothalamic amenorrhea; stress induced anovulation
MeSH Terms: conditions — Stress, Psychological | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavior therapy (Experimental): Cognitive behavior therapy consisting of 16 sessions over 20 weeks
  Interventions: Behavioral: Cognitive behavior therapy
- observation (Placebo Comparator): Subjects were called by telephone but were not given cognitive behavior therapy until the study phase was completed
  Interventions: Behavioral: Cognitive behavior therapy

INTERVENTIONS:
Behavioral: Cognitive behavior therapy — 16 sessions of 45 minutes each to review stress management

SUMMARY:
This is a randomized pilot study of the use of cognitive behavior therapy versus observation to treat functional hypothalamic amenorrhea, often termed stress-induced anovulation.

DETAILED DESCRIPTION:
The study enrollment was completed in 2003. The study results are being analyzed.

ELIGIBILITY:
Inclusion Criteria:

* women with functional hypothalamic amenorrhea
* day awake / night asleep schedule

Exclusion Criteria:

* eating disorders, depression, excessive exercise or any other cause of amenorrhea and anovulation other than functional hypothalamic amenorrhea
* weight loss greater than 10 pounds when amenorrhea developed
* running more than 10 miles per week or exercising more than 10 hours per week

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 1997-11; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
ovarian function | Change before and after 20 weeks of CBT or observation
  The change in ovarian function was assessed by comparing ovarian function before and after 20 weeks of CBT or observation using menses and serial estradiol and progesterone level as indices of ovarian function

SECONDARY OUTCOMES:
metabolism | Change before and after 20 weeks of CBT or observation
  The change in metabolism was assessed by measuring levels of cortisol, TSH, T4, free T4, T3, free T3, leptin in blood and by measuring weight before and after 20 weeks of CBT or observation

OTHER OUTCOMES:
psychological inventories | Change before and after 20 weeks of CBT or observation
  Attitudes were assessed before and after 20 weeks of CBT or observation using psychological inventories

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Berga, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Berga SL, Marcus MD, Loucks TL, Hlastala S, Ringham R, Krohn MA. Recovery of ovarian activity in women with functional hypothalamic amenorrhea who were treated with cognitive behavior therapy. Fertil Steril. 2003 Oct;80(4):976-81. doi: 10.1016/s0015-0282(03)01124-5. PMID 14556820
- [Derived] Kawwass JF, Sanders KM, Loucks TL, Rohan LC, Berga SL. Increased cerebrospinal fluid levels of GABA, testosterone and estradiol in women with polycystic ovary syndrome. Hum Reprod. 2017 Jul 1;32(7):1450-1456. doi: 10.1093/humrep/dex086. PMID 28453773
- [Derived] Michopoulos V, Mancini F, Loucks TL, Berga SL. Neuroendocrine recovery initiated by cognitive behavioral therapy in women with functional hypothalamic amenorrhea: a randomized, controlled trial. Fertil Steril. 2013 Jun;99(7):2084-91.e1. doi: 10.1016/j.fertnstert.2013.02.036. Epub 2013 Mar 16. PMID 23507474